CLINICAL TRIAL: NCT02832089
Title: Oral Carvedilol in Escalating Doses in the Acute Treatment of Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Andhra Medical College (Other Government)
Responsible Party: Principal Investigator, Ravi Venkatachelam Chitrapu, doctor, Andhra Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01AMCRVC
Record Dates: First submitted 2015-12-28; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; rate reduction
MeSH Terms: conditions — Atrial Fibrillation | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active arm (Experimental): single arm study with one group given oral carvedilol.
  Interventions: Drug: oral carvedilol

INTERVENTIONS:
Drug: oral carvedilol — oral carvedilol in escalating doses for reducing ventricular rate in AF patients
  Other Names: oral carvedilol in esclating doses

SUMMARY:
Oral carvedilol administered in escalating doses in patients with atrial fibrillation among patients with AF with fast ventricular rate.

DETAILED DESCRIPTION:
Patients with AF with FVR of any etiology were evaluated and given escalating doses of oral carvedilol in doses - 3.125mg OD, then 3.125 bid, then 6.25mg bid, then 12.5mg bid. The ECG was recorded regularly and analysed for rate reduction or control.

ELIGIBILITY:
Inclusion Criteria:

* AF with fast ventricular rate

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-12; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
reduction in ventricular rate in AF patients | 24 hours
  reduction in ventricular rate in patients with AF and fast ventricular rate.

IPD SHARING:
Plan to Share IPD: No